CLINICAL TRIAL: NCT03070288
Title: RGB(Red- Green-Blue) Measurement of the Nasal Mucosal Image: A New Diagnostic Parameter for Allergic Rhinitis
Brief Title: RGB(Red- Green-Blue) Measurement of the Nasal Mucosal Image
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Nazan Degirmenci, Principal Investigator, Bezmialem Vakif University
Other Study IDs: B.30.2.BAV.0.05.05/397
Record Dates: First submitted 2017-01-30; First posted 2017-03-03 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Allergic Rhinitis
Keywords: RGB; red-green-blue; rhinitis; allergic rhinitis; nasal mucosa
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Group 1: Red-green-blue measurements of nasal mucosa images of patients with allergic rhinitis
  Interventions: Other: Red-green-blue measurements of nasal mucosa image
- Group 2: Red-green-blue measurements of nasal mucosa images of normal healthy individuals
  Interventions: Other: Red-green-blue measurements of nasal mucosa image

INTERVENTIONS:
Other: Red-green-blue measurements of nasal mucosa image — Adobe Photoshop Elements 7.0 program automatically measures the numerical values of the RGB color components in the selected area

SUMMARY:
The aim of this study was to evaluate the color values of the nasal mucosa, which is easily assessable by a direct, non-invasive, objective photographic measurement, for the purpose of presenting a diagnostic objective parameter of allergic rhinitis (AR).

All patients and controls were examined by the same 4 mm 0⁰endoscope and light source, and all endoscopic photographs of the septum and both inferior turbinates were taken. Adobe Photoshop Elements 7.0 program was used to measure the numerical values of the red-green-blue (RGB) color components in endoscopic photographs of the nasal mucosa on the septum and inferior turbinates.

DETAILED DESCRIPTION:
This study enrolled 73 patients with AR (Group 1) and 73 normal healthy individuals(Group 2) with no nasal pathologies and respiratory tract infection attending to the outpatient clinic of the tertiary referral center. Patient's symptoms were questioned and noted by using Lebel Symptom Score Scale. Clinical examination was also done to help diagnose and exclude acute respiratory tract infection. All of the patients had positive skin prick test results for at least one of the most common aeroallergens. All patients and controls were examined by the same 4 mm 0⁰endoscope and light source, and all endoscopic photographs of the septum and both inferior turbinates were taken. Each image was marked with standardized points at the anterior part of the nasal mucosa on both sides (2 points each right and left sides of the anterior septum and 2 points each anterior part of the inferior turbinates). These points were numbered 1 and 2 over the right inferior turbinate; 3 and 4 over the right side of the anterior septum; 4 and 5 over the left inferior turbinate; 6 and 7 over the left side of the anterior septum. Adobe Photoshop Elements 7.0 program was used to measure the numerical values of the red-green-blue color components in endoscopic photographs of the nasal mucosa on the septum and inferior turbinates.

ELIGIBILITY:
Inclusion Criteria:

* Subject has positive skin prick test results
* Subject has more than 5 points of Lebel Symptom Score Scale
* Subjects between 18-60 ages
* Subjects with allergic rhinitis

Exclusion Criteria:

* Negative skin prick test results
* Acute respiratory tract infection existence
* Scores less than 5 points of Lebel Symptom Score Scale

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study enrolled 73 patients with allergic rhinitis (Group 1) and 73 normal healthy individuals(Group 2) with no nasal pathologies and respiratory tract infection attending to the outpatient clinic of the tertiary referral center. Patient's symptoms were questioned and noted by using Lebel Symptom Score Scale. Clinical examination was also done to help diagnose and exclude acute respiratory tract infection. All of the patients had positive skin prick test results for at least one of the most common aeroallergens.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
The difference of nasal mucosa color between groups | 3 months
  Nasal mucosa colors of the groups were measured with the numerical values of the RGB color components. All endoscopic photographs of the septum and both inferior turbinates of the patients and healthy individuals were taken while the examination at the outpatient clinic for three months. Adobe Photoshop Elements 7.0 program automatically measures the numerical values of the RGB color components in the pointed area. Color discoloration at the nasal mucosa of allergic patients compared with the healthy individuals by using RGB measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Degirmenci, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozturan O, Dogan R, Yenigun A, Veyseller B, Yildirim YS. Photographic Objective Alterations for Laryngopharyngeal Reflux Diagnosis. J Voice. 2017 Jan;31(1):78-85. doi: 10.1016/j.jvoice.2015.12.021. Epub 2016 Feb 9. PMID 26873421
- [Background] Tugrul S, Degirmenci N, Eren SB, Dogan R, Meric Hafiz A, Ozturan O. RGB measurements as a novel objective diagnostic test for otitis media with effusion. Acta Otolaryngol. 2015 Apr;135(4):342-7. doi: 10.3109/00016489.2014.984877. Epub 2015 Mar 5. PMID 25739969
- [Background] Osada T, Arakawa A, Sakamoto N, Ueyama H, Shibuya T, Ogihara T, Yao T, Watanabe S. Autofluorescence imaging endoscopy for identification and assessment of inflammatory ulcerative colitis. World J Gastroenterol. 2011 Dec 14;17(46):5110-6. doi: 10.3748/wjg.v17.i46.5110. PMID 22171146